CLINICAL TRIAL: NCT02930109
Title: A Phase I-II Study of Triciribine Phosphate Monohydrate (PTX-200) Plus Cytarabine in Refractory or Relapsed Acute Leukemia
Brief Title: A Study of PTX-200 (Triciribine) Plus Cytarabine in Refractory or Relapsed Acute Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prescient Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTX-200-AML-015
Record Dates: First submitted 2016-09-13; First posted 2016-10-12 (Estimated); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Acute Leukemia
MeSH Terms: interventions — Cytarabine

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- PTX-200 and cytarabine (Experimental): PTX-200 administered intravenously over 1 hour
  Phase I: 4 dose levels: 25 to 55 mg/m2 (with reduction to 15 mg/m2 if needed.
  Phase II: maximum tolerated dose. given as a 1 hour infusion
  Cytarabine administered by continuous infusion at a dose of 400 mg/m2/day for 4 days.
  Interventions: Drug: PTX-200; Drug: Cytarabine

INTERVENTIONS:
Drug: PTX-200 — During the Phase I study, increasing dose levels of PTX-200 will be administered as an intravenous infusion on Day 1 each cycle. Triciribine will be infused over 1 hour on Day 1 of each 21 day cycle. The initial dose level will be 25 mg/m2 and each dose level will be increased by 10 mg/m2 to a maximum dose of 55 mg/m2
  Other Names: Triciribine Phosphate Monohydrate
Drug: Cytarabine — Cytarabine will be given at a dose of 400 mg/m2 as a continuous IV infusion on days 3-7 of each cycle.
  Other Names: Ara-C

SUMMARY:
A phase I-II open label study of PTX-200 in combination with cytarabine in the treatment of relapsed or refractory acute leukemia.

DETAILED DESCRIPTION:
Study design: Phase I/II study The Phase I study is open-label with four increasing dose levels for up to four 21-day cycles. Safety and activity will be evaluated at the end of each cycle.

The Phase II study is open label with administration of the recommended phase dose of PTX-200 for up to four 21-day cycles. PTX-200 will be co-administered with cytarabine in both the Phase I and Phase II parts of the study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of the diagnosis of AML, ALL (acute lymphoblastic leukemia), or blast-phase CML (chronic myelogenous leukemia)
* Age ≥ 18 years
* ECOG Performance Status 0-2
* Patients must be able to give adequate informed consent

Exclusion Criteria:

* Hyperleukocytosis with ≥ 30,000 leukemic blasts/µL blood (hydroxyurea permitted up to 24 hours prior to beginning study drugs)
* Uncontrolled Disseminated Intravascular Coagulation (DIC)
* Uncontrolled diabetes mellitus
* Active, uncontrolled infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Treatment-related Adverse Events | 12 months
  Number of participants with treatment-related Adverse Events as assessed by CTCAE v4.0 that result in dose-limitations (Phase I)

SECONDARY OUTCOMES:
Phospho-Akt (pAkt) expression within CD34+ leukemic blasts | 12 months
  Change from baseline phospho-Akt (pAkt) signaling within CD34+ leukemic blasts and the ability of PTX-200 to downregulate p-Akt and its signaling at a variety of times

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lancet, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Cancer Center, Fairway, Kansas

IPD SHARING:
Plan to Share IPD: No